CLINICAL TRIAL: NCT03154164
Title: Study on the Learning Curve for Fundus First With Ultrasonic Tissue Coagulation in Elective Cholecystectomy
Acronym: LEFFE
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Other Study IDs: LEFFE
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Cholecystolithiasis
MeSH Terms: conditions — Cholecystolithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasonic tissue coagulation dissection — ultrasonic coagulation for dissection during laparoscopic cholecystectomy

SUMMARY:
The present study aims at analyzing the learning curve for fundus first with the ultrasonic tissue coagulation dissection technique in elective cholecystectomy. Patients included in the study are planned for an elective cholecystectomy, on the basis of the gallstone disease. All participating surgeons have experience of the traditional approach with electrocautery. The operation time as well as the surgeons own evaluation of difficulty and performance are noted. Selected films are analyzed by independent surgeons with experience of the fundus first technique. The Swedish registry of gallstone surgery and ERCP (GallRiks) are used to record the intra and postoperative complication rate.

DETAILED DESCRIPTION:
The present study aims at analyzing the learning curve for fundus first with the ultrasonic tissue coagulation dissection technique in elective cholecystectomy. Patients included in the study are planned for an elective cholecystectomy, on the basis of the gallstone disease. All participating surgeons have experience of the traditional approach with electrocautery, but limited experience from gallstone surgery with ultrasonic tissue coagulation dissection.

The operation time as well as the surgeons own evaluation of difficulty and performance are noted. Selected video recordings are analyzed by independent surgeons with experience of the fundus first technique. The Swedish registry of gallstone surgery and ERCP (GallRiks) are used to record the intra and postoperative complication rate. The study is intended to serve as a pilot study for a subsequent randomised controlled trial, comparing surgery with electrocautery and ultrasonic tissue coagulation dissection.

ELIGIBILITY:
Inclusion Criteria:

* Preoperatively discovered choledocholithiasis

Exclusion Criteria:

* Symptoms and signs of acute or chronic cholecystitis

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Dissection time | 6 hours
  Time required to dissect the gallbladder from the liver

SECONDARY OUTCOMES:
Level of technical complexity | 6 hours
  Level of technical complexity of the procedure assessed by the surgeon
Level of technical performance | 6 hours
  Level of technical performance during the procedure assessed by the surgeon
Technical performance | 6 hours
  Intraoperative technical performance assessed by an independent observer
Complication rate | 30 days
  Intra- and postoperative complication rate

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
All data will be saved and analysed after anonymising the participant.